CLINICAL TRIAL: NCT05568004
Title: The Effect of Different Exercise Types on Migraine Frequency in Individuals With Migraine :Randomized Controlled Study
Brief Title: The Effect of Different Exercise Types on Migraine Frequency in Individuals With Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Yunus Emre Meydanal, Resident physician of Sport Medicine Department, Ege University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 22-9T/12
Record Dates: First submitted 2022-09-27; First posted 2022-10-05 (Actual); Results first posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-02

CONDITIONS: Migraine; Chronic Migraine
Keywords: Headache; Exercise; Resistance exercises; Aerobic exercise
MeSH Terms: conditions — Migraine Disorders; Headache; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Combined exercise group (Experimental): Aerobic plus resistance exercise intervention
  Interventions: Behavioral: Combined exercise
- Aerobic exercise group (Experimental): Only aerobic exercise intervention
  Interventions: Behavioral: Aerobic exercise
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Combined exercise — aerobic plus resistance exercise
  Arms: Combined exercise group
Behavioral: Aerobic exercise — Only aerobic exercise
  Arms: Aerobic exercise group

SUMMARY:
The purpose of this study is to evaluate and compare the effect of different exercise types and combinations on migraine attacks in patients with migraine.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of migraine confirmed by a specialist neurologist according to International Classification of Headache Disorders, 3rd version(ICHD-3)
* Diagnosed as chronic migraine at the time of initial diagnosis (may have turned into episodic migraine under preventive treatment)
* At least 5 migraine attack/month in baseline diary
* No obstacle to exercise in the evaluation made with physical examination and ECG
* Diagnosed with migraine for at least 12 months
* Between the ages of 18-50

Exclusion Criteria:

* Exercising regularly in the last 6 months
* Presence of concomitant internal and neurological diseases
* Anti-psychotic drug use
* Drug, alcohol addiction
* Pregnancy, breastfeeding
* Patients who cannot reach the targeted exercise level

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-11-28 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yunus Emre Meydanal, Principal Investigator — Ege University Sport Medicine Clinic; Seckin Senısık, Study Director — Ege University Sport Medicine Clinic
Locations (1):
- Ege University Sport Medicine Clinic, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Headache Classification Committee of the International Headache Society (IHS) The International Classification of Headache Disorders, 3rd edition. Cephalalgia. 2018 Jan;38(1):1-211. doi: 10.1177/0333102417738202. No abstract available. PMID 29368949
- [Background] GBD 2015 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 310 diseases and injuries, 1990-2015: a systematic analysis for the Global Burden of Disease Study 2015. Lancet. 2016 Oct 8;388(10053):1545-1602. doi: 10.1016/S0140-6736(16)31678-6. PMID 27733282
- [Background] GBD 2015 Neurological Disorders Collaborator Group. Global, regional, and national burden of neurological disorders during 1990-2015: a systematic analysis for the Global Burden of Disease Study 2015. Lancet Neurol. 2017 Nov;16(11):877-897. doi: 10.1016/S1474-4422(17)30299-5. Epub 2017 Sep 17. PMID 28931491
- [Background] Lipton RB, Bigal ME, Diamond M, Freitag F, Reed ML, Stewart WF; AMPP Advisory Group. Migraine prevalence, disease burden, and the need for preventive therapy. Neurology. 2007 Jan 30;68(5):343-9. doi: 10.1212/01.wnl.0000252808.97649.21. PMID 17261680
- [Background] Ertas M, Baykan B, Orhan EK, Zarifoglu M, Karli N, Saip S, Onal AE, Siva A. One-year prevalence and the impact of migraine and tension-type headache in Turkey: a nationwide home-based study in adults. J Headache Pain. 2012 Mar;13(2):147-57. doi: 10.1007/s10194-011-0414-5. Epub 2012 Jan 14. PMID 22246025
- [Background] Calhoun AH, Ford S, Millen C, Finkel AG, Truong Y, Nie Y. The prevalence of neck pain in migraine. Headache. 2010 Sep;50(8):1273-7. doi: 10.1111/j.1526-4610.2009.01608.x. Epub 2010 Jan 18. PMID 20100298
- [Background] Lipton RB, Silberstein SD. Episodic and chronic migraine headache: breaking down barriers to optimal treatment and prevention. Headache. 2015 Mar;55 Suppl 2:103-22; quiz 123-6. doi: 10.1111/head.12505_2. PMID 25662743
- [Background] Smitherman TA, Burch R, Sheikh H, Loder E. The prevalence, impact, and treatment of migraine and severe headaches in the United States: a review of statistics from national surveillance studies. Headache. 2013 Mar;53(3):427-36. doi: 10.1111/head.12074. Epub 2013 Mar 7. PMID 23470015
- [Background] Buse DC, Manack AN, Fanning KM, Serrano D, Reed ML, Turkel CC, Lipton RB. Chronic migraine prevalence, disability, and sociodemographic factors: results from the American Migraine Prevalence and Prevention Study. Headache. 2012 Nov-Dec;52(10):1456-70. doi: 10.1111/j.1526-4610.2012.02223.x. Epub 2012 Jul 25. PMID 22830411
- [Background] Stewart WF, Ricci JA, Chee E, Morganstein D, Lipton R. Lost productive time and cost due to common pain conditions in the US workforce. JAMA. 2003 Nov 12;290(18):2443-54. doi: 10.1001/jama.290.18.2443. PMID 14612481
- [Background] Blumenfeld AM, Varon SF, Wilcox TK, Buse DC, Kawata AK, Manack A, Goadsby PJ, Lipton RB. Disability, HRQoL and resource use among chronic and episodic migraineurs: results from the International Burden of Migraine Study (IBMS). Cephalalgia. 2011 Feb;31(3):301-15. doi: 10.1177/0333102410381145. Epub 2010 Sep 2. PMID 20813784
- [Background] Lipton RB, Stewart WF, Sawyer J, Edmeads JG. Clinical utility of an instrument assessing migraine disability: the Migraine Disability Assessment (MIDAS) questionnaire. Headache. 2001 Oct;41(9):854-61. PMID 11703471
- [Background] Lipton RB, Bigal ME, Stewart WF. Clinical trials of acute treatments for migraine including multiple attack studies of pain, disability, and health-related quality of life. Neurology. 2005 Dec 29;65(12 Suppl 4):S50-8. doi: 10.1212/wnl.65.12_suppl_4.s50. PMID 16385104
- [Background] Buse DC, Manack A, Serrano D, Turkel C, Lipton RB. Sociodemographic and comorbidity profiles of chronic migraine and episodic migraine sufferers. J Neurol Neurosurg Psychiatry. 2010 Apr;81(4):428-32. doi: 10.1136/jnnp.2009.192492. Epub 2010 Feb 17. PMID 20164501
- [Background] Bigal ME, Serrano D, Reed M, Lipton RB. Chronic migraine in the population: burden, diagnosis, and satisfaction with treatment. Neurology. 2008 Aug 19;71(8):559-66. doi: 10.1212/01.wnl.0000323925.29520.e7. PMID 18711108
- [Background] Giannini G, Cevoli S, Sambati L, Cortelli P. Migraine: risk factor and comorbidity. Neurol Sci. 2012 May;33 Suppl 1:S37-41. doi: 10.1007/s10072-012-1029-6. PMID 22644168
- [Background] Stewart WF, Wood GC, Manack A, Varon SF, Buse DC, Lipton RB. Employment and work impact of chronic migraine and episodic migraine. J Occup Environ Med. 2010 Jan;52(1):8-14. doi: 10.1097/JOM.0b013e3181c1dc56. PMID 20042889
- [Background] Negro A, D'Alonzo L, Martelletti P. Chronic migraine: comorbidities, risk factors, and rehabilitation. Intern Emerg Med. 2010 Oct;5 Suppl 1:S13-9. doi: 10.1007/s11739-010-0457-7. PMID 20865469
- [Background] Wang SJ, Chen PK, Fuh JL. Comorbidities of migraine. Front Neurol. 2010 Aug 23;1:16. doi: 10.3389/fneur.2010.00016. eCollection 2010. PMID 21188255
- [Background] Antonaci F, Nappi G, Galli F, Manzoni GC, Calabresi P, Costa A. Migraine and psychiatric comorbidity: a review of clinical findings. J Headache Pain. 2011 Apr;12(2):115-25. doi: 10.1007/s10194-010-0282-4. Epub 2011 Jan 6. PMID 21210177
- [Background] Breslau N. Psychiatric comorbidity in migraine. Cephalalgia. 1998 Aug;18 Suppl 22:56-8; discussion 58-61. doi: 10.1177/0333102498018s2210. No abstract available. PMID 9793713
- [Background] Ashina S, Serrano D, Lipton RB, Maizels M, Manack AN, Turkel CC, Reed ML, Buse DC. Depression and risk of transformation of episodic to chronic migraine. J Headache Pain. 2012 Nov;13(8):615-24. doi: 10.1007/s10194-012-0479-9. Epub 2012 Sep 25. PMID 23007859
- [Background] McWilliams LA, Goodwin RD, Cox BJ. Depression and anxiety associated with three pain conditions: results from a nationally representative sample. Pain. 2004 Sep;111(1-2):77-83. doi: 10.1016/j.pain.2004.06.002. PMID 15327811
- [Background] Lucchetti G, Peres MF, Lucchetti AL, Mercante JP, Guendler VZ, Zukerman E. Generalized anxiety disorder, subthreshold anxiety and anxiety symptoms in primary headache. Psychiatry Clin Neurosci. 2013 Jan;67(1):41-9. doi: 10.1111/j.1440-1819.2012.02405.x. PMID 23331287
- [Background] Chen YC, Tang CH, Ng K, Wang SJ. Comorbidity profiles of chronic migraine sufferers in a national database in Taiwan. J Headache Pain. 2012 Jun;13(4):311-9. doi: 10.1007/s10194-012-0447-4. Epub 2012 Apr 12. PMID 22527034
- [Background] Queiroz LP, Peres MF, Piovesan EJ, Kowacs F, Ciciarelli MC, Souza JA, Zukerman E. A nationwide population-based study of migraine in Brazil. Cephalalgia. 2009 Jun;29(6):642-9. doi: 10.1111/j.1468-2982.2008.01782.x. Epub 2009 Feb 2. PMID 19187337
- [Background] Varkey E, Hagen K, Zwart JA, Linde M. Physical activity and headache: results from the Nord-Trondelag Health Study (HUNT). Cephalalgia. 2008 Dec;28(12):1292-7. doi: 10.1111/j.1468-2982.2008.01678.x. Epub 2008 Sep 11. PMID 18771495
- [Background] Wober C, Brannath W, Schmidt K, Kapitan M, Rudel E, Wessely P, Wober-Bingol C; PAMINA Study Group. Prospective analysis of factors related to migraine attacks: the PAMINA study. Cephalalgia. 2007 Apr;27(4):304-14. doi: 10.1111/j.1468-2982.2007.01279.x. PMID 17376107
- [Background] Koseoglu E, Akboyraz A, Soyuer A, Ersoy AO. Aerobic exercise and plasma beta endorphin levels in patients with migrainous headache without aura. Cephalalgia. 2003 Dec;23(10):972-6. doi: 10.1046/j.1468-2982.2003.00624.x. PMID 14984230
- [Background] Varkey E, Cider A, Carlsson J, Linde M. A study to evaluate the feasibility of an aerobic exercise program in patients with migraine. Headache. 2009 Apr;49(4):563-70. doi: 10.1111/j.1526-4610.2008.01231.x. Epub 2008 Sep 9. PMID 18783448
- [Background] Varkey E, Cider A, Carlsson J, Linde M. Exercise as migraine prophylaxis: a randomized study using relaxation and topiramate as controls. Cephalalgia. 2011 Oct;31(14):1428-38. doi: 10.1177/0333102411419681. Epub 2011 Sep 2. PMID 21890526
- [Background] Domingues RB, Teixeira AL, Domingues SA. Physical practice is associated with less functional disability in medical students with migraine. Arq Neuropsiquiatr. 2011 Feb;69(1):39-43. doi: 10.1590/s0004-282x2011000100009. PMID 21359421
- [Background] Kroll LS, Hammarlund CS, Linde M, Gard G, Jensen RH. The effects of aerobic exercise for persons with migraine and co-existing tension-type headache and neck pain. A randomized, controlled, clinical trial. Cephalalgia. 2018 Oct;38(12):1805-1816. doi: 10.1177/0333102417752119. Epub 2018 Jan 15. PMID 29333870
- [Background] Hanssen H, Minghetti A, Magon S, Rossmeissl A, Rasenack M, Papadopoulou A, Klenk C, Faude O, Zahner L, Sprenger T, Donath L. Effects of different endurance exercise modalities on migraine days and cerebrovascular health in episodic migraineurs: A randomized controlled trial. Scand J Med Sci Sports. 2018 Mar;28(3):1103-1112. doi: 10.1111/sms.13023. Epub 2018 Jan 8. PMID 29161767
- [Background] Darabaneanu S, Overath CH, Rubin D, Luthje S, Sye W, Niederberger U, Gerber WD, Weisser B. Aerobic exercise as a therapy option for migraine: a pilot study. Int J Sports Med. 2011 Jun;32(6):455-60. doi: 10.1055/s-0030-1269928. Epub 2011 Apr 6. PMID 21472632
- [Background] Lemmens J, De Pauw J, Van Soom T, Michiels S, Versijpt J, van Breda E, Castien R, De Hertogh W. The effect of aerobic exercise on the number of migraine days, duration and pain intensity in migraine: a systematic literature review and meta-analysis. J Headache Pain. 2019 Feb 14;20(1):16. doi: 10.1186/s10194-019-0961-8. PMID 30764753
- [Background] Garber CE, Blissmer B, Deschenes MR, Franklin BA, Lamonte MJ, Lee IM, Nieman DC, Swain DP; American College of Sports Medicine. American College of Sports Medicine position stand. Quantity and quality of exercise for developing and maintaining cardiorespiratory, musculoskeletal, and neuromotor fitness in apparently healthy adults: guidance for prescribing exercise. Med Sci Sports Exerc. 2011 Jul;43(7):1334-59. doi: 10.1249/MSS.0b013e318213fefb. PMID 21694556
- [Background] Irby MB, Bond DS, Lipton RB, Nicklas B, Houle TT, Penzien DB. Aerobic Exercise for Reducing Migraine Burden: Mechanisms, Markers, and Models of Change Processes. Headache. 2016 Feb;56(2):357-69. doi: 10.1111/head.12738. Epub 2015 Dec 8. PMID 26643584
- [Background] Misra UK, Kalita J, Tripathi GM, Bhoi SK. Is beta endorphin related to migraine headache and its relief? Cephalalgia. 2013 Apr;33(5):316-22. doi: 10.1177/0333102412473372. Epub 2013 Jan 11. PMID 23314782
- [Background] Beavers KM, Brinkley TE, Nicklas BJ. Effect of exercise training on chronic inflammation. Clin Chim Acta. 2010 Jun 3;411(11-12):785-93. doi: 10.1016/j.cca.2010.02.069. Epub 2010 Feb 25. PMID 20188719
- [Background] Dietrich A, McDaniel WF. Endocannabinoids and exercise. Br J Sports Med. 2004 Oct;38(5):536-41. doi: 10.1136/bjsm.2004.011718. PMID 15388533
- [Background] Hoffman MD, Hoffman DR. Does aerobic exercise improve pain perception and mood? A review of the evidence related to healthy and chronic pain subjects. Curr Pain Headache Rep. 2007 Apr;11(2):93-7. doi: 10.1007/s11916-007-0004-z. PMID 17367586
- [Background] Houle TT, Butschek RA, Turner DP, Smitherman TA, Rains JC, Penzien DB. Stress and sleep duration predict headache severity in chronic headache sufferers. Pain. 2012 Dec;153(12):2432-2440. doi: 10.1016/j.pain.2012.08.014. Epub 2012 Oct 13. PMID 23073072
- [Background] John PJ, Sharma N, Sharma CM, Kankane A. Effectiveness of yoga therapy in the treatment of migraine without aura: a randomized controlled trial. Headache. 2007 May;47(5):654-61. doi: 10.1111/j.1526-4610.2007.00789.x. PMID 17501846
- [Background] Andersen CH, Jensen RH, Dalager T, Zebis MK, Sjogaard G, Andersen LL. Effect of resistance training on headache symptoms in adults: Secondary analysis of a RCT. Musculoskelet Sci Pract. 2017 Dec;32:38-43. doi: 10.1016/j.msksp.2017.08.003. Epub 2017 Aug 14. PMID 28854396
- [Background] Sullivan AB, Scheman J, Venesy D, Davin S. The role of exercise and types of exercise in the rehabilitation of chronic pain: specific or nonspecific benefits. Curr Pain Headache Rep. 2012 Apr;16(2):153-61. doi: 10.1007/s11916-012-0245-3. PMID 22258395
- [Background] Hagen K, Einarsen C, Zwart JA, Svebak S, Bovim G. The co-occurrence of headache and musculoskeletal symptoms amongst 51 050 adults in Norway. Eur J Neurol. 2002 Sep;9(5):527-33. doi: 10.1046/j.1468-1331.2002.00451.x. PMID 12220386
- [Background] Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-81. PMID 7154893
- [Background] Skinner JS, Hutsler R, Bergsteinova V, Buskirk ER. The validity and reliability of a rating scale of perceived exertion. Med Sci Sports. 1973 Summer;5(2):94-6. No abstract available. PMID 4721013
- [Background] Lamb KL, Eston RG, Corns D. Reliability of ratings of perceived exertion during progressive treadmill exercise. Br J Sports Med. 1999 Oct;33(5):336-9. doi: 10.1136/bjsm.33.5.336. PMID 10522637
- [Background] Muyor JM. Exercise Intensity and Validity of the Ratings of Perceived Exertion (Borg and OMNI Scales) in an Indoor Cycling Session. J Hum Kinet. 2013 Dec 31;39:93-101. doi: 10.2478/hukin-2013-0072. eCollection 2013 Dec 18. PMID 24511345
- [Background] Colado JC, Garcia-Masso X, Triplett TN, Flandez J, Borreani S, Tella V. Concurrent validation of the OMNI-resistance exercise scale of perceived exertion with Thera-band resistance bands. J Strength Cond Res. 2012 Nov;26(11):3018-24. doi: 10.1519/JSC.0b013e318245c0c9. PMID 22210471
- [Background] ASTRAND PO, RYHMING I. A nomogram for calculation of aerobic capacity (physical fitness) from pulse rate during sub-maximal work. J Appl Physiol. 1954 Sep;7(2):218-21. doi: 10.1152/jappl.1954.7.2.218. No abstract available. PMID 13211501

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who applied to Ege University Hospital Neurology Department of Headache policlinic were recruited based on neurology physician up to International Headache Disorder Classification 3rd version (ICHD-3). Participants were enrolled to study between November 2022- January 2024.
Pre-assignment Details: Of 32 enrolled participants , 24 participants filled out baseline headache diaries regularly and were randomized to groups
Groups:
- Combined Exercise Group: Aerobic plus resistance exercise intervention
  Combined exercise: aerobic plus resistance exercise For 12 weeks participants did aerobic exercise 3 times a week. One session took 45 minutes During this time patients did five different resistance exercise with elastic bands three times a week. Participants started resistance exercises with 2 sets of 8 repetitions, with a gradual increase until 3 sets of 12 repetitions were reached at the end of the first month.
- Aerobic Exercise Group: Only aerobic exercise intervention
  Aerobic exercise: Only aerobic exercise For 12 weeks participants did aerobic exercise 3 times a week. One session took 45 minutes
- Control Group: no intervention
Period: Overall Study
Arm/Group | Combined Exercise Group | Aerobic Exercise Group | Control Group
Started | 8 | 8 | 8
Completed | 8 | 8 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Combined Exercise Group | Aerobic Exercise Group | Control Group | Total
Number analyzed (Participants) | 8 | 8 | 8 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 39 (13) | 36 (11) | 44 (5) | 39.8 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 8 | 22
  Male | 2 | 0 | 0 | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body weight [Mean (Standard Deviation); unit: kilogram] | 74 (14) | 68 (10) | 75 (12) | 71.9 (12.12)
Height [Mean (Standard Deviation); unit: centimeter] | 166 (10) | 163 (5) | 162 (2) | 163.5 (6.35)
Body mass index [Mean (Standard Deviation); unit: kilogram/square meter] | 26.60 (3.46) | 25.50 (3.84) | 28.45 (5.15) | 26.85 (4.21)
Migraine duration [Mean (Standard Deviation); unit: years] | 13.2 (12.9) | 8.5 (10) | 16.8 (7.8) | 12.8 (10.5)
Number of Participants with Migraine Aura [Count of Participants; unit: Participants] — Number of participants in that group with migraine headache accompanied by aura (determined using participants' baseline diaries)
  Participants | 2 | 1 | 1 | 4
Preventive drugs number [Mean (Standard Deviation); unit: mean number of medication used] — Numbers indicate the mean number of preventive drug used in the baseline period before the intervention in this group.
  mean number of medication used | 1 (1) | 1 (1) | 1 (0) | 1 (0.48)
Beta blocker use [Count of Participants; unit: Participants] — The numbers show how many patients in that group used this type of medication in the baseline period before the intervention
  Participants | 4 | 5 | 6 | 15
Serotonin and norepinephrine reuptake inhibitors (SNRIs) use [Count of Participants; unit: Participants] — The numbers show how many patients in that group used this type of medication in the baseline period before the intervention
  Participants | 5 | 2 | 3 | 10
Tricyclic antidepressants (TCAs) [Count of Participants; unit: Participants] — The numbers show how many patients in that group used this type of medication in the baseline period before the intervention
  Participants | 2 | 1 | 0 | 3
Number of participants using medication for migraine attack treatment(triptan) [Number; unit: participants] — The numbers show how many patients in that group used this type of medication(triptan) in the baseline period before the intervention (In our study, all participants using preventive drugs for migraine were using a single type of medication, triptan.)
  participants | 5 | 7 | 7 | 19

OUTCOME MEASURES:

1. Primary Outcome: Change in the Number of Days With Migraine (in Migraine Frequency)
Description: Defined as the number of days with a migraine headache in a month
Time Frame: Baseline and Week 12 and Week 20
Population: all participants who were assigned to the arm
Measure: Mean (Standard Deviation); unit: days/month
Arm/Group | Combined Exercise Group | Aerobic Exercise Group | Control Group
Number analyzed (Participants) | 8 | 8 | 8
days/month
  Baseline | 9.9 (4.2) | 12.4 (4.5) | 11.8 (3.4)
  End of 12 weeks(Post intervention) | 6.3 (3.4) | 8 (4.5) | 10.6 (2.3)
  End of 8 weeks (follow up) | 6.5 (3.4) | 8.8 (4.1) | 10.6 (3.2)
Statistical Analysis 1: Comparison: Combined Exercise Group; Test type: Superiority; p = 0.001, ANOVA — A p-value of < 0.05 was considered statistically significant for all analyses.Two-tailed testing was used in nature of hypothesis testing; p value for change over time within the group, Friedman 2-way ANOVA test was applied; Statistical analysis was conducted by a researcher using the Statistical Package for Social Sciences (SPSS) version 26.0. The Shapiro-Wilk test and histograms evaluated the data for normal distribution, and the Levene test confirmed homogeneous variances between groups (p > 0.05). Continuous data following a normal distribution are presented as mean ± standard deviation (SD). The independent samples t test or Mann-Whitney U test was used to compare independent continuous data between groups, while the chi-square or Fisher's exact test was used to compare categorical data. Friedman two-way ANOVA was used to analyze dependent variables, while the two-way mixed ANOVA was used to examine the changes between groups over time. Before the two-way mixed ANOVA, boxplot evaluation confirmed no outliers. Mauchly's sphericity test showed that the assumption of sphericity for two-way interaction was met. Tukey's correction was used for pairwise subgroup comparisons
Statistical Analysis 2: Comparison: Aerobic Exercise Group; A p-value of < 0.05 was considered statistically significant for all analyses.Two-tailed testing was used in nature of hypothesis testing; Test type: Superiority; p = 0.001, ANOVA; p value for change over time within the group, Friedman 2-way ANOVA test was applied
Statistical Analysis 3: Comparison: Control Group; Test type: Superiority; p = 0.166, ANOVA — [p-value comment as in outcome 1, analysis 1]; p value for change over time within the group, Friedman 2-way ANOVA test was applied

2. Secondary Outcome: Average Intensity of Headache
Description: A categorical, 11 points visual analogue scale will be used to rate each headache between 0-10. Higher scores mean higher severity headache
Time Frame: Baseline and Week 12 and Week 20
Population: all participants who were assigned to the arm
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: headaches
Arm/Group | Combined Exercise Group | Aerobic Exercise Group | Control Group
Number analyzed (Participants) | 8 | 8 | 8
Number analyzed (headaches) | 43 | 47 | 44
score on a scale
  Baseline | 7 (0.9) | 7.5 (1.2) | 7.4 (0.5)
  Week 12(Post intervention) | 6.3 (1.2) | 6.8 (1) | 7 (0.9)
  Week 20(follow up) | 6.6 (0.9) | 6.6 (1.1) | 7.1 (0.8)
Statistical Analysis 1: Comparison: Combined Exercise Group; Statistical Package for Social Sciences (SPSS) 26.0 package program was used to analyze the data. The suitability of normal distribution of the data was evaluated with Shapiro Wilk and histograms. Numerical data complying with normal distribution are presented as mean±standard deviation (SD). . Friedman 2-way ANOVA was used to analyze dependent variables. Two-way mixed ANOVA test was used to examine the changes between groups over time; Test type: Superiority; p = 0.074, ANOVA — [p-value comment as in outcome 1, analysis 1]; p value for change over time within the group, Friedman 2-way ANOVA test was applied
Statistical Analysis 2: Comparison: Aerobic Exercise Group; Test type: Superiority — A p-value of < 0.05 was considered statistically significant for all analyses.Two-tailed testing was used in nature of hypothesis testing; p = 0.074, ANOVA; p value for change over time within the group, Friedman 2-way ANOVA test was applied
Statistical Analysis 3: Comparison: Control Group; Test type: Superiority; p = 0.311, ANOVA — A p-value of < 0.05 was considered statistically significant for all analyses; p value for change over time within the group, Friedman 2-way ANOVA test was applied

3. Secondary Outcome: Anxiety
Description: Hospital Anxiety and Depression Scale (HADS) will be used. Score could score between 0 and 21 for either anxiety or depression subscale . Higher points are associated with worse anxiety or depression
Time Frame: Baseline and Week 12 and Week 20
Population: all participants who were assigned to the arm
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Exercise Group | Aerobic Exercise Group | Control Group
Number analyzed (Participants) | 8 | 8 | 8
score on a scale
  Baseline | 10.3 (3.5) | 7.8 (3.9) | 6.3 (3.9)
  Week 12 (post intervention) | 8.5 (2.6) | 6 (2.6) | 6.3 (3.3)
  Week 20 (follow up) | 8.3 (2.4) | 6.5 (2.4) | 5.8 (3.4)
Statistical Analysis 1: Comparison: Combined Exercise Group; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.018, ANOVA — A p-value of < 0.05 was considered statistically significant for all analyses; *p-value for changes over time within the group; Friedman's two-way ANOVA test was applied
Statistical Analysis 2: Comparison: Aerobic Exercise Group; Test type: Superiority; p = 0.152, ANOVA — A p-value of < 0.05 was considered statistically significant for all analyses; *p-value for changes over time within the group; Friedman's two-way ANOVA test was applied
Statistical Analysis 3: Comparison: Control Group; Test type: Superiority; p = 0.438, ANOVA — A p-value of < 0.05 was considered statistically significant for all analyses; *p-value for changes over time within the group; Friedman's two-way ANOVA test was applied

4. Secondary Outcome: Depression
Description: Hospital Anxiety and Depression Scale (HADS) will be used. Score could score between 0 and 21 for either anxiety or depression subscales . Higher points are associated with worse anxiety or depression
Time Frame: Baseline and Week 12 and Week 20
Population: all participants who were assigned to the arm
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Exercise Group | Aerobic Exercise Group | Control Group
Number analyzed (Participants) | 8 | 8 | 8
score on a scale
  Baseline | 7 (5.8) | 6.8 (3.1) | 5.4 (2.8)
  Week 12 (post intervention) | 5.6 (4.4) | 5.8 (2.9) | 4.9 (2.1)
  Week 20 (follow up) | 5.5 (4.3) | 6.1 (3.3) | 5.3 (1.9)
Statistical Analysis 1: Comparison: Combined Exercise Group; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.135, ANOVA — A p-value of < 0.05 was considered statistically significant for all analyses; *p-value for changes over time within the group; Friedman's two-way ANOVA test was applied
Statistical Analysis 2: Comparison: Aerobic Exercise Group; Test type: Superiority; p = 0.203, ANOVA — A p-value of < 0.05 was considered statistically significant for all analyses; *p-value for changes over time within the group; Friedman's two-way ANOVA test was applied
Statistical Analysis 3: Comparison: Control Group; Test type: Superiority; p = 0.593, ANOVA — A p-value of < 0.05 was considered statistically significant for all analyses; *p-value for changes over time within the group; Friedman's two-way ANOVA test was applied

5. Secondary Outcome: Migraine Specific Quality of Life
Description: Migraine Disability Assessment (MIDAS) questionnaire will be used . There is no upper or lower limit on scoring. More than 21 points show severe disability. Higher points mean more disability.MIDAS Grade/ MIDAS Score: Little or No Disability 0-5 , Mild Disability 6-10 , Moderate Disability 11-20 , Severe Disability 21+
Time Frame: Baseline and Week 12 and Week 20
Population: all participants who were assigned to the arm
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Exercise Group | Aerobic Exercise Group | Control Group
Number analyzed (Participants) | 8 | 8 | 8
score on a scale
  Baseline | 49 (17.8) | 46.8 (37) | 42.8 (23.1)
  Week 12 (post intervention) | 32.1 (14.8) | 30.6 (25.2) | 39.5 (19.3)
  Week 20 (follow up) | 35.1 (15.4) | 32.4 (26.4) | 40 (19.7)
Statistical Analysis 1: Comparison: Combined Exercise Group; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.001, ANOVA — A p-value of < 0.05 was considered statistically significant for all analyses; *p-value for changes over time within the group; Friedman's two-way ANOVA test was applied
Statistical Analysis 2: Comparison: Aerobic Exercise Group; Test type: Superiority; p = 0.021, ANOVA — A p-value of < 0.05 was considered statistically significant for all analyses; *p-value for changes over time within the group; Friedman's two-way ANOVA test was applied
Statistical Analysis 3: Comparison: Control Group; Test type: Superiority; p = 0.081, ANOVA — A p-value of < 0.05 was considered statistically significant for all analyses; *p-value for changes over time within the group; Friedman's two-way ANOVA test was applied

6. Secondary Outcome: Aerobic Capacity Measurement V02 Max
Description: Astrand submaximal bicycle ergometer test will be used to measure aerobic capacity.
Time Frame: Baseline and Week 12 and Week 20
Population: all participants who were assigned to the arm
Measure: Mean (Standard Deviation); unit: mililiter/kilogram/minute
Arm/Group | Combined Exercise Group | Aerobic Exercise Group | Control Group
Number analyzed (Participants) | 8 | 8 | 8
mililiter/kilogram/minute
  Baseline | 30.1 (3) | 29.5 (2.1) | 28 (1.6)
  Week 12 (post intervention) | 33.4 (3.8) | 32.5 (2.2) | 28.1 (1.7)
  Week 20 (follow up) | 32.1 (3.6) | 31.1 (2) | 28.1 (1.9)
Statistical Analysis 1: Comparison: Combined Exercise Group; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.001, ANOVA — A p-value of < 0.05 was considered statistically significant for all analyses; *p-value for changes over time within the group; Friedman's two-way ANOVA test was applied
Statistical Analysis 2: Comparison: Aerobic Exercise Group; Test type: Superiority; p < 0.001, ANOVA — A p-value of < 0.05 was considered statistically significant for all analyses; *p-value for changes over time within the group; Friedman's two-way ANOVA test was applied
Statistical Analysis 3: Comparison: Control Group; Test type: Superiority; p = 0.747, ANOVA — A p-value of < 0.05 was considered statistically significant for all analyses; *p-value for changes over time within the group; Friedman's two-way ANOVA test was applied

7. Secondary Outcome: Change in Physical Activity Level
Description: The International Physical Activity Questionnaires (IPAQ) short form will be used. Scoring is not classical numerical type. For activity type and duration are important for scoring. Higher points means more physical activity
Time Frame: Baseline and Week 12 and Week 20
Population: all participants who were assigned to the arm
Measure: Mean (Standard Deviation); unit: metabolic equivalent /week
Arm/Group | Combined Exercise Group | Aerobic Exercise Group | Control Group
Number analyzed (Participants) | 8 | 8 | 8
metabolic equivalent /week
  Baseline | 565.1 (328.9) | 585.1 (427.9) | 415.1 (272.9)
  Week 12 (post intervention) | 1338.4 (156.3) | 1542.4 (379.9) | 660.8 (514.6)
  Week 20 (follow up) | 854.8 (301.7) | 867 (438.5) | 552.1 (359.7)
Statistical Analysis 1: Comparison: Combined Exercise Group; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.001, ANOVA — A p-value of < 0.05 was considered statistically significant for all analyses; *p-value for changes over time within the group; Friedman's two-way ANOVA test was applied
Statistical Analysis 2: Comparison: Aerobic Exercise Group; Test type: Superiority; p < 0.001, ANOVA — A p-value of < 0.05 was considered statistically significant for all analyses; p-value for changes over time within the group; Friedman's two-way ANOVA test was applied
Statistical Analysis 3: Comparison: Control Group; Test type: Superiority; p = 0.05, ANOVA — A p-value of < 0.05 was considered statistically significant for all analyses; p-value for changes over time within the group; Friedman's two-way ANOVA test was applied

ADVERSE EVENTS:
Time Frame: 20 weeks
Arm/Group | Combined Exercise Group | Aerobic Exercise Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8

LIMITATIONS AND CAVEATS:
Low sample size Performing exercises without supervision Not having a group that does only resistance exercise Participants continue their current preventive medications without changing the dose during the intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2025-02-15): https://cdn.clinicaltrials.gov/large-docs/04/NCT05568004/Prot_001.pdf
  • Statistical Analysis Plan (2024-06-16): https://cdn.clinicaltrials.gov/large-docs/04/NCT05568004/SAP_002.pdf